CLINICAL TRIAL: NCT05148182
Title: Metabolomics Characterization of Biomarkers of ASCVD and Prediction Model
Acronym: MEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Other Study IDs: MEAL
Record Dates: First submitted 2021-11-05; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Atherosclerosis; Prediction Model
Keywords: metabolomics; Atherosclerosis; Biomarkers; prediction model
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The instrument platforms of gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS) are used to metabonomic analysis. Small molecular metabolites in blood were measured by LC-MS and GC-MS.The instrument platforms of GC-MS and LC-MS are used. The samples tested on GC-MS platform need to be derivatized, mainly for the detection of polar and weak polar metabolites with molecular weight not higher than 1000Da and low boiling point; LC-MS uses different liquid phase systems to detect polar and weak polar metabolites, lipids and lipid soluble metabolites respectively; The same sample needs to be detected through five data acquisition modes on three mass spectrometry platforms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low risk: According to the China PAR equations and Chinese guidelines and consensus on cardiovascular risk assessment and management, it is considered as low-risk population.
- medium risk: According to the China PAR equations and Chinese guidelines and consensus on cardiovascular risk assessment and management, it is considered as medium-risk population.
- high risk: According to the China PAR equations and Chinese guidelines and consensus on cardiovascular risk assessment and management, it is considered as high-risk population.

SUMMARY:
1. Describe the risk factors and metabonomics characteristics of atherosclerotic cardiovascular disease in Chinese patients.
2. Establish accurate prediction model of atherosclerotic heart disease.

DETAILED DESCRIPTION:
According to the Chinese cardiovascular disease report released in 2017, cardiovascular disease death is the leading cause of death of urban and rural residents, so cardiovascular disease risk assessment is particularly important. The development of cardiovascular risk assessment model was dated from Framingham Heart Study which first proposed the concept of risk factors, and then adjusted the model several times. In 2016, the China-PAR evaluated the cardiovascular disease risk of Chinese population. However, the application of metabolomics in coronary heart disease is a rapidly developing field and also a new field .

Therefore, the aim of this study was to

1.Describe the risk factors of atherosclerotic cardiovascular disease and the characteristics of metabolomics in Chinese population.

2. Establish an accurate prediction model of atherosclerotic heart disease. Research plan：

1. 1869 risk-stratified people were recruited.
2. Plasma samples were collected incluing disease status and other potential influencing factors.
3. Through the high-throughput detection of body metabolites, combined with multivariate statistical analysis, the metabolic markers with significant difference in different risk levels were screened for risk prediction.
4. All recruited people underwent coronary angiography.
5. The distribution of age and gender in each group should be matched and balanced as far as possible.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the population is 18 or more than 18 years old.
2. According to China PAR equations, Chinese guidelines and consensus on cardiovascular risk assessment and management，it is considered as healthy, low, medium, high and extremely high risk group.
3. The subjects read and fully understood the patient's instructions and signed the informed consent

Exclusion Criteria:

1. Refused to sign informed consent.
2. ACS is caused by surgery, trauma, or other diseases.
3. Age less than 18 years old.
4. Pregnant women.
5. In the past 3 months, the patients were treated with trauma surgery.
6. There are aortic dissection, pulmonary embolism, pneumonia, pericarditis, myocarditis, stress cardiomyopathy.
7. Severe heart failure.
8. Liver and kidney failure.
9. Blood borne infectious diseases: including HIV / AIDS, hepatitis B, hepatitis C, etc.
10. Patients with a history of malignancies, autoimmune diseases, severe infectious diseases and trauma.
11. Any condition (such as travel, speech disorder, mental disorder) that the researcher believes can significantly limit the completion of the patient's follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to China PAR equations and Chinese guidelines and consensus on cardiovascular risk assessment and management, the patients were defined as low, medium, high risk groups.
Sampling Method: Probability Sample
Enrollment: 1869 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Metabolomics Characterization of Biomarkers | 3 years
  Metabonomics analysis uses a non targeted detection method to detect polar compounds and lipid compounds in blood. The characteristic peaks of substances that can be detected are detected by chromatography Series platform, and then these characteristic peaks are compared with the standard library containing more than 8000 metabolites to annotate the compounds and screen out the differential metabolites between groups.
Coronary vascularization. | 3 years
  Coronary vascularization includes percutaneous coronary intervention, or/and percutaneous coronary artery dilatation, or/and percutaneous coronary artery bypass grafting.
All cause mortality | 3 years
  which refers to the total death caused by various causes in a certain period.
Cardiac mortality | 3 years
  Cardiac death refers to the death caused by serious cardiac dysfunction or failure which caused by heart disease or injury in a certain period.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Cardiology,Shanghai Tenth People's Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai